CLINICAL TRIAL: NCT07200336
Title: Efficacy of Anti-IL-5 Therapy Combined With Simple Polypectomy Versus Extended Endoscopic Sinus Surgery in Patients With CRSwNP: A Multicenter Randomized Controlled Trial
Brief Title: Anti-IL-5 Therapy With Simple Polypectomy Versus Extended Endoscopic Sinus Surgery for CRSwNP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Huabin Li, Professor and Director of the Department of Allergy Center, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPESS-2025
Record Dates: First submitted 2025-09-13; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Keywords: Anti-IL-5; Biologic-Surgical Combination; Extended Sinus Surgery; SNOT-22; Type 2 Inflammation; Recurrence
MeSH Terms: conditions — Recurrence | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anti-IL-5 Monotherapy (Experimental): Mepolizumab 100mg subcutaneously every 4 weeks for 24 weeks
  Interventions: Drug: Mepolizumab
- Anti-IL-5 + Simple Polypectomy (Experimental): Combined therapy: A 100 mg dose of mepolizumab is initiated subcutaneously 2 weeks after simple polypectomy. Mepolizumab will be administered subcutaneously every 4 weeks for 24 weeks.
  Interventions: Drug: Mepolizumab; Procedure: Simple Polypectomy
- Anti-IL-5 + Extended Endoscopic Sinus Surgery (Experimental): Combined therapy: A 100 mg dose of mepolizumab is initiated subcutaneously 2 weeks after Extended Endoscopic Sinus Surgery. Mepolizumab will be administered subcutaneously every 4 weeks for 24 weeks.
  Interventions: Drug: Mepolizumab; Procedure: Extended Endoscopic Sinus Surgery

INTERVENTIONS:
Drug: Mepolizumab — Subcutaneous injection of mepolizumab is administered every 4 weeks for a total treatment duration of 24 weeks.
Procedure: Simple Polypectomy — Removal of nasal polyps in the middle meatus and superior turbinate region via the middle meatus and olfactory cleft, without opening the involved sinuses and without resection of diseased bone.
  Arms: Anti-IL-5 + Simple Polypectomy
Procedure: Extended Endoscopic Sinus Surgery — 1. Complete opening of all sinuses
  2. Resection of diseased mucosa and hyperplastic bone
  3. Ethmoid skeletonization with middle turbinectomy
  4. Draf IIb/III frontal dissection when indicated by CT severity.
  Arms: Anti-IL-5 + Extended Endoscopic Sinus Surgery

SUMMARY:
This study compares two surgical approaches combined with anti-IL-5 therapy in patients with chronic rhinosinusitis with nasal polyps (CRSwNP). Patients will be randomly assigned to one of the three groups: (1) anti-IL-5 alone, (2) anti-IL-5 with simple polyp removal, or (3) anti-IL-5 with extended sinus surgery. The aim of this study is to see if a less invasive surgery (simple polyp removal) with anti-IL-5 works as well as more extensive surgery with anti-IL-5. Participants will be followed for 1 to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Endoscopy shows bilateral nasal polyps, with bilateral NPS ≥4 (≥2 per side)
2. Nasal obstruction symptoms >3 months, nasal obstruction score ≥2 (total 3 points) and/or hyposmia ≥2 (maximum 3 points)
3. Evidence of type 2 inflammation: Nasal polyp tissue Eos >55/HPF or >27% of inflammatory cells; or Peripheral blood Eos ≥6.9% (without asthma) or ≥3.7% (with asthma) Note: Meet any 2 of the above 3 criteria
4. Failure after 4 weeks of standard medical therapy including: Intranasal corticosteroids >4 weeks; Other agents (oral steroids, macrolides, antihistamines, leukotriene receptor antagonists, decongestants, antibiotics) permitted as needed

Exclusion Criteria:

1. Cystic fibrosis, Young's syndrome, Kartagener syndrome, antrochoanal polyp, or rhinitis medicamentosa
2. Acute upper respiratory infection within 2 weeks
3. Asthma exacerbation within 1 month
4. HIV infection
5. Parasitic infection within 6 months
6. History of hypersensitivity to investigational drugs (except aspirin intolerance)
7. Hypersensitivity to monoclonal antibodies or anti-IL-5 agents
8. Oral steroid therapy within 1 month
9. Pregnancy planning, current pregnancy, or lactation
10. Uncontrolled systemic diseases
11. Have a history of previous sinus surgery for CRSwNP
12. Significant septal deviation affecting unilateral ventilation (mild deviation allowed)
13. Investigator judgment of unsuitability for cohort study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2029-10-10 (Estimated); Study Completion 2031-10-10 (Estimated)

PRIMARY OUTCOMES:
The Change in SNOT-22 Score | Baseline,Month12
  The 22-item Sinonasal Outcome Test (SNOT-22) is a questionnaire comprising 22 questions on health-related quality of life in rhinosinusitis. For each item, patients provide a subjective rating on a scale from 0 to 5, where 0 represents "No problem" and 5 represents "Problem as bad as it can be." The total score is the sum of all items and ranges from a minimum of 0 to a maximum of 110. A higher total score indicates a worse outcome, reflecting a poorer quality of life due to rhinosinusitis.
Change in Nasal Congestion Score | Baseline, Month 12
  The Nasal Congestion Score (NCS) is a patient-reported outcome measure that assesses the subjective severity of nasal congestion. The score ranges from a minimum of 0 to a maximum of 3, where 0 represents "No nasal congestion" and 3 represents "The most severe nasal congestion." A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Change in SNOT-22 Score | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,24,36 month after biological treatment initiation
  The 22-item Sinonasal Outcome Test (SNOT-22) is a questionnaire comprising 22 questions on health-related quality of life in rhinosinusitis. For each item, patients provide a subjective rating on a scale from 0 to 5, where 0 represents "No problem" and 5 represents "Problem as bad as it can be." The total score is the sum of all items and ranges from a minimum of 0 to a maximum of 110. A higher total score indicates a worse outcome, reflecting a poorer quality of life due to rhinosinusitis.
Change in Nasal Congestion Score | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,24,36 month after biological treatment initiation
  The Nasal Congestion Score (NCS) is a patient-reported outcome measure that assesses the subjective severity of nasal congestion. The score ranges from a minimum of 0 to a maximum of 3, where 0 represents "No nasal congestion" and 3 represents "The most severe nasal congestion." A higher score indicates a worse outcome.
Change in Nasal Polyp Score (NPS) | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,12,24,36 month after biological treatment initiation
  The Nasal Polyp Score (NPS) is an objective assessment tool, evaluated by a clinician, used to grade the size of nasal polyps. Each nasal cavity is scored separately on a scale from 0 to 4. The total score is the sum of the scores from both nostrils and ranges from a minimum of 0 to a maximum of 8. A higher score indicates larger nasal polyps and a worse outcome. The scoring criteria are as follows:
  0: No polyps.
  1. Small polyps in the middle meatus.
  2. Polyps in the middle meatus reaching below the inferior border of the middle turbinate.
  3. Large polyps reaching beyond the inferior border of the middle turbinate or with medial extension from the middle turbinate.
  4. Polyps completely obstructing the nasal cavity.
Change in Modified Lund-Kennedy Score | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,12,24,36 month after biological treatment initiation
  The modified Lund-Kennedy (MLK) score is an objective endoscopic evaluation performed by a clinician. A higher score indicates a worse outcome. It scores nasal polyps, edema, and discharge (0-2 for each) per nostril. The total score ranges from 0 to 12, with a higher score indicating worse endoscopic status.
Change in Blood Eosinophil percentage | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,12,24,36 month after biological treatment initiation
Change in Lund-Mackay CT Score | Baseline, at 6,12, 24,36 month after biological treatment
  The Lund-Mackay CT scoring system is an objective radiological assessment. It evaluates the extent of opacification on sinus computed tomography (CT) scans in six anatomical regions per side: anterior ethmoid sinuses, posterior ethmoid sinuses, maxillary sinuses, sphenoid sinuses, frontal sinuses, and the ostiomeatal complex. Each region is scored from 0 (no abnormality) to 2 (complete opacification). The total score, which is the sum of scores from all regions across both sides, ranges from a minimum of 0 to a maximum of 24. A higher total score indicates greater disease severity.
Change in Olfactory Function | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,12,24,36 month after biological treatment initiation
  We will provide patients with an olfactory questionnaire, asking them to respond to the following questions. Each question will have a corresponding score: 0 points for "strongly disagree," 1 point for "partially agree," 2 points for "incompletely agree," and 3 points for "strongly agree."
  The questions include:
  I feel my sense of smell has become much worse than before. Compared to before the onset of olfactory dysfunction, the taste of food has changed.
  Sometimes I can smell unpleasant odors that others cannot detect. Some pleasant smells that others enjoy are unpleasant to me. My biggest issue is that, compared to before the onset of olfactory dysfunction, smells are perceived differently.
  Due to changes in my sense of smell, I dine out less often than before. I worry that I will not be able to adapt to the changes in my sense of smell in the future.
  Due to changes in my sense of smell, I feel more anxious than before. Changes in my sense of smell often make me feel angry.
Change in FeNO and nNO | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 3,6,12,24,36 month after first biological treatment
Need for Systemic Corticosteroid | 2 Weeks after first treatment(operation or biologic treatment) ,at 1,2,3,4,5,6,12,24,36 month after biological treatment initiation
Objective Olfactory function Test | Baseline, 2 Weeks after first treatment(operation or biologic treatment) ,at 3,6,12,24,36 month after biological treatment initiation
  Olfactory function was evaluated by the Sniffin' Sticks test, containing olfactory threshold (T), discrimination (D) and identification (I) tests . Score for the threshold test range between 1 and 16, while the scores of the other two tests range between 0 and 16. The results of the three tests were calculated as a total TDI score (range 1- 48), which was used to define functional anosmia (TDI ≤ 16), hyposmia (16 < TDI < 31), or normosmia (TDI ≥ 31). If the patients had only been assessed by the identification test, the I score was used to define functional anosmia (I ≤ 8), hyposmia (8 < I ≤ 11), or 113 normosmia (I > 11).

CONTACTS AND LOCATIONS:
Overall Officials: Huabin Li, PhD, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (17):
- China (17):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Longgang District Central Hospital of Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - Affiliated Hangzhou First People's Hospital,School of Medicine, Westlake University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subspecialty Group of Rhinology, Editorial Board of Chinese Journal of Otorhinolaryngology Head and Neck Surgery; Subspecialty Group of Rhinology, Society of Otorhinolaryngology Head and Neck Surgery, Chinese Medical Association. [Guideline for diagnosis and treatment of chronic rhinosinusitis (2024)]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2025 Mar 7;60(3):221-249. doi: 10.3760/cma.j.cn115330-20250116-00051. No abstract available. Chinese. PMID 40147886
- [Background] Han JK, Bachert C, Fokkens W, Desrosiers M, Wagenmann M, Lee SE, Smith SG, Martin N, Mayer B, Yancey SW, Sousa AR, Chan R, Hopkins C; SYNAPSE study investigators. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Oct;9(10):1141-1153. doi: 10.1016/S2213-2600(21)00097-7. Epub 2021 Apr 16. PMID 33872587
- [Background] Homoe AS, Aanaes K, Tidemandsen JE, Holbaek HC, Niclas R, Badsberg SG, Holmegaard LBI, Backer V. Superior Benefits of Combining Mepolizumab With Sinus Surgery Compared to Mepolizumab Alone: Results From a Randomised 6-Month Trial. Int Forum Allergy Rhinol. 2025 Jul;15(7):724-733. doi: 10.1002/alr.23562. Epub 2025 Mar 10. PMID 40065601
- [Background] Maza-Solano J, Callejon-Leblic A, Martin-Jimenez D, Moreno-Luna R, Gonzalez-Garcia J, Cuvillo A, Sanchez-Gomez S. Omalizumab Treatment in Uncontrolled Asthma and CRSwNP Patients, with Previous Endoscopic Sinus Surgery, to Improve Quality of Life and Endoscopic Outcomes: a Two-Year Real-Life Study. Curr Allergy Asthma Rep. 2023 Oct;23(10):555-566. doi: 10.1007/s11882-023-01106-w. Epub 2023 Aug 30. PMID 37644255
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Xian M, Yan B, Song X, Chen J, Tang J, Jiang Y, Wan L, Liu W, Xue J, Cao Z, Yu Y, Yang X, Shi L, Wang G, Xu Y, Yang Y, Ye J, Jiang L, Quan F, Tan G, Liu F, Xu Z, Zhang X, Li J, Su L, Yang Y, Fan J, He G, Zhu L, Wang X, Wang M, Shen S, Li J, Li H, Wei X, Yu H, Liu Z, Ma R, Liu H, Liu J, Lv W, Yang Q, Zhu D, Cheng L, Wang C, Zhang L. Chinese Position Paper on Biologic Therapy for Chronic Rhinosinusitis With Nasal Polyps. Allergy. 2025 May;80(5):1208-1225. doi: 10.1111/all.16519. Epub 2025 Mar 5. PMID 40042059